CLINICAL TRIAL: NCT01696344
Title: Does AF Termination Without Additional Ablation Influence Outcome?
Brief Title: Does Atrial Fibrillation (AF) Termination Without Additional Ablation Influence Outcome?
Acronym: TARGET
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: California Pacific Medical Center (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, TCAI, Texas Cardiac Arrhythmia Research Foundation
Other Study IDs: TCAI_TARGET
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: LSPAF; AF termination; PVAI; nonPV triggers; Long-standing persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: No additional ablation after AF termination(PVAI only)
  Interventions: Procedure: PVAI
- Cohort 2: Additional ablation of extra-PV triggers before and after isoproterenol-challenge after AF termination (PVAI + ablation of extra-PV triggers)
  Interventions: Procedure: PVAI + ablation of extraPV triggers

INTERVENTIONS:
Procedure: PVAI
  Other Names: Pulmonary vein antrum isolation
  Groups: Cohort 1
Procedure: PVAI + ablation of extraPV triggers — PVAI followed by ablation of extra-PV triggers originating from sites other than pulmonary veins such as superior vena cava, ligament of Marshall, coronary sinus, crista terminalis, left atrial (LA) posterior wall and LA appendage
  Groups: Cohort 2

SUMMARY:
This prospective study aims to investigate if termination of atrial fibrillation (AF) after pulmonary vein antrum isolation (PVAI) without additional ablation of non-PV triggers, in long-standing persistent (LSP) AF, is enough to ensure long-term success.

DETAILED DESCRIPTION:
Background: AF is a heterogeneous arrhythmia. At its simplest, it is triggered by rapidly firing foci around pulmonary veins (PV) and can be cured by isolation of PV alone. Evidences suggest that when high frequency of atrial activation is maintained for relatively longer period (as in persistent or long-standing AF), ion channel remodeling changes the electrophysiologic substrate and lead to AF permanence. Therefore, PVAI alone, as anticipated, demonstrates to have limited success rate in persistent and LSP AF and additional ablations beyond PVAI involving substrate modification are advocated by many experts in electrophysiology. However, there is yet no consensus on the ablation strategy for long-standing AF. It is still not clear whether AF termination during ablation could be considered as an ablation endpoint or not, as earlier studies have reported results that are at variance with each other. Some studies have suggested that termination of AF during ablation is associated with reduced recurrence of arrhythmia while others detected no association of AF termination with long-term maintenance of sinus rhythm (SR) in persistent or LSP-AF.Therefore this study aims to examine ablation outcomes in LSP-AF patients with AF termination with or without additional ablation of extra-PV triggers.

Hypothesis: AF termination does not eliminate the need for additional ablations in achieving long-term ablation success in LSP-AF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. LSP-AF patients experiencing AF termination during ablation
3. Ability to understand and provide signed informed consent

Exclusion Criteria:

1. Previous left atrial catheter ablation or MAZE procedure in left atrium
2. Reversible causes of atrial arrhythmia such as hyperthyroidism, sarcoidosis, pulmonary embolism etc

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Drug-refractory long-standing persistent atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
AF recurrence | 3 years
  Any episode of AF/AT longer than 30 seconds will be considered as recurrence. Episodes that occur during the first 3 months of the procedure (blanking period) will not be considered as recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — TCAI
Locations (2):
- United States (2):
  - St. david's Medical Center, Austin, Texas
  - Texas Cardiac arrhythmia Institute, St. David's Hospital, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided